CLINICAL TRIAL: NCT06496191
Title: FMT for Alcohol Use Disorder in Cirrhotics: A Randomized Controlled Trial.
Brief Title: FMT for Alcohol Use Disorder in Cirrhotics.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-FMT-03
Record Dates: First submitted 2024-06-14; First posted 2024-07-11 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-06

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT + SMT (Experimental): Therapy with Fecal microbiota transplantation with SMT (Baclofen + AUD counselling). - Single dose (30gm/90ml) of FMT will be given via upper GI gastroduodenoscope at D4.
  Interventions: Biological: FMT; Other: SMT
- Placebo + SMT (Active Comparator): Placebo therapy with SMT (Baclofen + AUD counselling)
  Interventions: Other: SMT; Other: Placebo

INTERVENTIONS:
Biological: FMT — - Single dose (30gm/90ml) of FMT will be given via upper GI gastroduodenoscope at D4
  Arms: FMT + SMT
Other: SMT — Baclofen + AUD counselling
Other: Placebo — Placebo identical to the FMT arm.
  Arms: Placebo + SMT

SUMMARY:
* Title "FMT for Alcohol Use Disorder in cirrhotics: A Randomized Controlled Trial"
* The aim of the study is to study the efficacy of Fecal microbiota transplantation in patients with Alcohol liver disease over a 6 month duration without liver related side effects. The project will be conducted at ILBS over the period of 1 year.
* The concept is to test the efficacy of FMT in alcohol related cirrhotics by its effect on achieving and maintaining abstinence and in reducing lapses and relapses. Thereby reducing the progression of alcoholic liver disease as continued ethanol consumption is an important predictor in increasing overall morbidity and mortality.

DETAILED DESCRIPTION:
Hypothesis :- - FMT is useful in reducing craving and return to heavy drinking in patients with alcohol related cirrhosis with active drinking, through modulation of gut microbiota and correction of dysbiosis

Aim and Objective -

- To assess the efficacy of FMT in decreasing lapse, relapses and maintaining alcohol abstinence in AUD in patients with cirrhosis

Study population:

- Patients with cirrhosis with recent alcohol use attending outpatient clinic at ILBS, New Delhi

Study design:

- Open label, parallel group, randomized, controlled study.

Study period:

- 1 year

Sample size with justification:

- Assuming that abstinence in Placebo group is 50% and we assume that there will be 40% absolute increase in FMT group (90%; Bajaj JS, Hepatology 2021) with alpha 5 and power of 80%, investigator need to enroll 48 cases, further assuming 10 % dropout rate it was decided to enroll 54 cases that is 27 in each group.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive patients with alcohol related cirrhosis with serum bilirubin <5mg/dl with an active alcohol consumption atleast within last 4 weeks aged between 18 -70yrs.
2. Fulfilling DSM - 5 criteria for alcohol use disorder (Association, 2013).

Exclusion Criteria:

1. Pregnancy
2. Acute illness or fever on the day of planned FMT
3. Ongoing/Past 2 weeks antibiotic use
4. Unclear diagnosis of CLD
5. Non-elective hospitalization within last month
6. Serum bilirubin >5mg/dl
7. Grade 2 or more Ascites
8. Any Episode of HE Grade 2 or more or requiring hospital admission within 3 months
9. Episode of AVB within last 3 months
10. Treatment with corticosteroids/Immunosupression within the past 60 days
11. Unwilling to participate
12. Dependence on any other substance (except Nicotine)
13. Psychiatric disorder requiring pharmacotherapy/Suicidal tendency
14. Known untreated, in-situ luminal GI cancers & chronic intrinsic GI diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving and maintaining alcohol abstinence at 4 weeks | 4 weeks

SECONDARY OUTCOMES:
Gut microbiome alterations and relative abundance of gut associated bacteria. | 12 weeks
  Gut microbiome composition will be assessed by 16s Metagenomics
Proportion of patients who got FMT at 12 weeks without liver related adverse effects compared to placebo. | 12 weeks
Proportion of patients maintaining abstinence from alcohol at 3 & 6 months. | 3 and 6 months
Craving measures will be assessed based on pre-existing structured and validated questionnaires (Obsessive Compulsive Drinking Scale (OCDS) and Visual Analog Scale (VAS). | 4,12 weeks and 6 months
  VAS ranges from 0 to 10, where 0 means no craving and 10 means most craving or strongest drive to consume alcohol, in our thesis)
Proportion of patients developing lapse and relapse at 4,12 weeks and 6 months. | 4,12 weeks and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India